CLINICAL TRIAL: NCT01422590
Title: Pharmacodynamics After Concomitant Administration With Mitiglinide and Sitagliptin Compared to Mitiglinide, Sitagliptin Single Administration in Patients With Type 2 Diabetes
Brief Title: Pharmacodynamics of Mitiglinide/Sitagliptin Compared to Mitiglinide and Sitagliptin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-04-071
Record Dates: First submitted 2011-08-10; First posted 2011-08-24 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: sitagliptin; mitiglinide; type 2 diabetes mellitus; Pharmacodynamics; Safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; mitiglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin
- Mitiglinide (Active Comparator)
  Interventions: Drug: Mitiglinide
- Sitagliptin + Mitiglinide (Experimental)
  Interventions: Drug: Sitagliptin, Mitiglinide

INTERVENTIONS:
Drug: Sitagliptin — Single oral administration of sitagliptin 100 mg
  Arms: Sitagliptin
Drug: Mitiglinide — Single oral administration of mitiglinide 10 mg
  Arms: Mitiglinide
Drug: Sitagliptin, Mitiglinide — Concomitant administration of sitagliptin 100 mg and mitiglinide 10 mg
  Arms: Sitagliptin + Mitiglinide

SUMMARY:
1. Explore pharmacodynamics

   * glucose
   * insulin
   * C-peptide
   * glucagon
   * intact GLP-1
   * DPP-4 activity
   * CGMS (continuous glucose monitoring system)
2. Assess Safety

   * adverse events
   * clinical laboratory test
   * physical examination

DETAILED DESCRIPTION:
Pharmacodynamic assessment

* CGMS data is obtained from day 1 to day 3 (48 hours)
* PD is measured before (day 1) and after drug administration (day 2)

  1. AUC of glucose, insulin, C-peptide, glucagon, intact GLP-1, DPP-4 activity
  2. MAGE (mean amplitude of glycemic excursion) from CGMS data

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with type 2 diabetes mellitus
* 6.5% ≤ HbA1c < 9.0%
* Stopped treatment of sulfonylurea and biguanide for more than 8 weeks
* Stopped treatment of other anti-diabetic agents for more than 12 weeks
* 16 kg/m2 ≤ body mass index < 30 kg/m2

Exclusion Criteria:

* Fasting glucose ≥ 200 mg/dL
* Required insulin therapy
* Patients with neuropathy, retinopathy or renopathy
* Contraindicated for mitiglinide or sitagliptin

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve) of plasma glucose | day 1 and day 2 of each period
  Differences of AUC before treatment (day 1) and after treatment (day 2) is compared between treatment groups
AUC of insulin | day 1 and day 2 of each period
  Differences of AUC before treatment (day 1) and after treatment (day 2) is compared between treatment groups
AUC of intact GLP-1 | day 1 and day 2 of each period
  Differences of AUC before treatment (day 1) and after treatment (day 2) is compared between treatment groups
AUC of C-peptide | day 1 and day 2 of each period
  Differences of AUC before treatment (day 1) and after treatment (day 2) is compared between treatment groups
AUC of glucagon | day 1 and day 2 of each period
  Differences of AUC before treatment (day 1) and after treatment (day 2) is compared between treatment groups
MAGE | day 1 and day 2 of each period
  Differences of MAGE before treatment (day 1) and after treatment (day 2) is compared between treatment groups
AUC of DPP-4 activity | day 1 and day 2 of each period
  Differences of AUC before treatment (day 1) and after treatment (day 2) is compared between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Hur, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jung JA, Kaku K, Kim JH, Kim JR, Ko JW, Lee SY, Huh W. Additive postprandial glucose-lowering effects of mitiglinide and sitagliptin in patients with type 2 diabetes mellitus. Adv Ther. 2013 Nov;30(11):1018-29. doi: 10.1007/s12325-013-0072-x. Epub 2013 Nov 19. PMID 24249434